CLINICAL TRIAL: NCT02322424
Title: Predictive Risk Factors for Pancreatic Fistula Grade C After Pancreaticoduodenectomy: Prospective Large Observational Study
Brief Title: Predictive Risk Factors for Pancreatic Fistula Grade C After Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University
Other Study IDs: Japan-Taiwan PD Project
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Disease of Pancreatic Head or Periampullary Lesions to Require Pancreaticoduodenectomy
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients who undergo pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy

SUMMARY:
Pancreatic fistula (PF) grade C, defined by the International Study Group of Pancreatic Fistula (ISGPF) is associated with a life-threatening complication after pancreaticoduodenectomy(PD). Therefore, The aim of this study is to clarify the risk factors for grade C PF by Japan and Taiwan cooperative project.

DETAILED DESCRIPTION:
Pancreatic fistula (PF) grade C, defined by the International Study Group of Pancreatic Fistula (ISGPF) is associated with a life-threatening complication after pancreaticoduodenectomy(PD). The rate of grade C PF has been reported 2.5-6%, however, it is critical complication after PD. A large number of enrolled patients will be needed to clarify the risk factors for grade C PF. Therefore, this study design is prospective large observational study at multi-center in Japan and Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Disease of pancreatic head or periampullary lesions to require pancreaticoduodenectomy
2. Age: 20 years or older
3. PS (ECOG performance status scale) 0-1 at the time of enrollment
4. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. patients with severe respiratory disorder required oxygen inhalation
2. patients with severe liver dysfunction
3. patients with chronic renal failure with dialysis
4. patients who are unfit for this study as determined by the attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3,000 patients who undergo pancreaticoduodenectomy (PD) in Japan and Taiwan
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula grade C | 90 days after pancreaticoduodenectomy

SECONDARY OUTCOMES:
Incidence of overall pancreatic fistula (grade A, grade B and grade C) | 90 days after pancreaticoduodenectomy
Incidence of clinical relevant pancreatic fistula (grade B and grade C) | 90 days after pancreaticoduodenectomy
Incidence of postpancreatecomy hemorrhage(PPH) | 90 days after pancreaticoduodenectomy
Cut-off value of drain amylase fluid on POD1 to distinguish pancreatic fistula grade C with grade A and grade B | 90 days after pancreaticoduodenectomy
Cut-off value of drain amylase fluid on POD1 to distinguish pancreatic fistula grade B and C with grade A | 90 days after pancreaticoduodenectomy
Morbidity | 90 days after pancreaticoduodenectomy
30-day mortality | 30 days after pancreaticoduodenectomy
90-day mortality | 90 days after pancreaticoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, M.D., PhD., Principal Investigator — Wakayama Medical University
Locations (1):
- Chang Gun Memorial Hospital, Linkou District, Taiwan